CLINICAL TRIAL: NCT05131009
Title: Differences in Incidence and Risk Factors of Postoperative Pulmonary Complications Between Patients Undergoing Abdominal Surgery in Plateau and Plain Areas
Brief Title: Postoperative Pulmonary Complications Between Patients Undergoing Abdominal Surgery in Plateau and Plain Areas
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Qinghai People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PPC202108
Record Dates: First submitted 2021-10-25; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Postoperative Pulmonary Complications;Abdominal Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with pulmonary complications following abdominal surgery
- Patients without pulmonary complications following abdominal surgery

SUMMARY:
This study aims to collect perioperative diagnosis and treatment information of patients undergoing abdominal surgery at plateau and plain areas , collect blood and others samples for laboratory testing when necessary, analyzing the data to clarify the incidence and risk factors of pulmonary complications in patients undergoing abdominal surgery at different altitudes, so as to reduce the risk of pulmonary complications and even death in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old；
2. scheduled for elective abdominal surgery under general anesthesia；
3. ASAⅠ-Ⅲ

Exclusion Criteria:

1. Patients and their family members refused to be enrolled；
2. patients were unable to communicate because of language disorders such as dementia and hearing impairment；
3. patients were admitted to ICU 48 hours before operation；
4. preoperative diagnosis of ARDS, aspiration pneumonia, pulmonary embolism or pulmonary edema or other acute respiratory diseases；
5. mechanical ventilation within one week before operation；
6. death or discharge within 24 hours after operation；
7. second operation due to postoperative complications

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older who planned elective abdominal surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
incidence and risk factors of pulmonary complications | 1 week after surgery

SECONDARY OUTCOMES:
ventilation duration,length of stay in ICU and Hospital Stay and death | within the 30 days after surgery
incidence of Major Extrapulmonary Complications | within the 30 days after surgery
Biomarkers | 1 week after surgery
incidence and risk factors of various specific pulmonary complications | 1 week after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China